CLINICAL TRIAL: NCT02733744
Title: A Pilot Study to Determine the Feasibility of Fecal MicrobiotaTransplantation (FMT) in Hematopoietic Stem Cell Transplantation (HSCT) Recipients
Brief Title: Fecal Microbiota Transplantation After HSCT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Yi-Bin A. Chen, MD, MD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-023
Record Dates: First submitted 2016-03-30; First posted 2016-04-11 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Bone Marrow Transplantation
Keywords: Stem cell transplant; fecal microbiota transplantation
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fecal Microbiota Transplant (Experimental): Each participant will undergo allogeneic hematopoietic stem cell transplantation, according to institutional standards.
  Participants will receive a single standard dose of oral Fecal Microbiota Transplantation (FMT), which is 15 capsules per day for two consecutive days, for a total of 30 capsules. Participants will be asked to fast for 4 hours prior to and 1 hour following capsule intake. Capsules will be individually handed to participants by a research nurse or physician. Each capsule will be taken with a sip of water.
  Interventions: Biological: Fecal Microbiota Transplantation (FMT)

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation (FMT) — FMT will be given through the ingestion of 30 capsules (15 capsules daily x 2 consecutive days)
  Other Names: FMT

SUMMARY:
This research study is studying an intervention called fecal microbiota transplantation (FMT). Patients who are scheduled to undergo Hematopoietic Stem Cell Transplantation are invited to take part in this clinical trial to undergo empiric FMT soon after hematopoietic engraftment. The primary endpoint will be to assess the feasibility of FMT in this population and to assess safety.

DETAILED DESCRIPTION:
The microbiome (spectrum of bacteria in a patient's gut) is thought to play a role in helping to shape one's immune system given its direct contact with normal cells in our intestine. Recent studies have suggested that a microbiome with very few bacteria (low diversity) seems to be bad for health and a high-diversity microbiome (many different species) appears to be good. This appears to be true even for patients after HSCT where low diversity microbiome status has correlated with infections, GVHD and overall survival.

Fecal microbiota transplantation (FMT) is routinely performed for an infection caused by Clostridium difficile but is not yet approved by the FDA as a treatment for any disease. FMT restores a high diversity microbiome. It is hoped that through FMT, overall outcomes after HSCT can potentially be improved.

FMT will be performed in the first 3 weeks after recovery of white blood cells after HSCT. The source of FMT will be from healthy 3rd party donors. FMT will be performed through the ingestion of 30 capsules over 2 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 18 and ≤ 65 years old
* Patients designated to undergo myeloablative or intermediate intensity allogeneic peripheral blood or bone marrow hematopoietic cell transplantation. Consent will be obtained prior to admission for HSCT. Patients receiving any donor source of stem cells are eligible. Eligible conditioning regimens are those defined as myeloablative by Consensus Criteria (Bacigalupo 2009) as well as the combination of fludarabine with melphalan (100-140 mg/mg2)
* Any Graft-vs-Host disease (GVHD) prophylaxis regimen is allowed.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%, see Appendix A)
* Patients with adequate physical function as measured by

  * Cardiac: Left ventricular ejection fraction at rest must be ≥ 40%, or shortening fraction >25%.
  * Hepatic:

    * Bilirubin ≤ 2.5 mg/dL, except for patients with Gilbert's syndrome or hemolysis
    * Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and Alkaline Phosphatase < 5 x Upper Limit of Institutional Normal Range (ULN).
  * Renal: Serum creatinine within normal range, or if serum creatinine is outside normal range, then renal function (measured or estimated creatinine clearance or GFR) ≥ 40millileters/min/1.73m2.
  * Pulmonary: Diffusing lung capacity for carbon monoxide (DLCO) (corrected for hemoglobin), Forced expiratory volume in 1 second (FEV1) and Forced vital capacity (FVC) ≥ 50% predicted.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study and for 3 months after FMT.
* Ability to understand and the willingness to sign a written informed consent document, including the willingness to accept risk of unrelated donor stool.
* Ability to swallow oral medications.

Exclusion Criteria:

* Prior allogeneic hematopoietic stem cell transplantation. (Patients may have received a prior autologous hematopoietic stem cell transplant.)
* Participants who are receiving any other investigational agents.
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with active or uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
* Patients with history of primary idiopathic myelofibrosis or any severe marrow fibrosis.
* Planned use of prophylactic donor lymphocyte infusion (DLI) therapy.
* Delayed gastric emptying syndrome
* Known chronic aspiration
* Patients with a history of significant allergy to foods not excluded from the donor diet (excluded foods are tree nuts, peanuts, shellfish, eggs)
* Pregnant and breast-feeding women are ineligible because they are not eligible for hematopoietic stem cell transplantation.
* HIV-positive participants are ineligible.
* Participants who are unable to swallow pills.
* Participants with end-stage liver disease (cirrhosis)
* Participants with acute, active gastrointestinal infection (e.g., typhlitis, diverticulitis, appendicitis)
* Participants with inflammatory bowel disease (e.g., ulcerative colitis, Crohn's)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-05; Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Feasibility measured by number of participants able to ingest 15 FMT capsules over a 2-day period | 2 days
  Number of participants able to ingest 15 FMT capsules over a 2 day period.

SECONDARY OUTCOMES:
Progression Free Survival | 2 years
Overall Survival | 2 years
Cumulative Incidence Of aGVHD | 2 years
Non-Relapse Mortality Rate | 2 years
Number of participants with treatment-related adverse events | 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Bin Chen, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts general Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DeFilipp Z, Peled JU, Li S, Mahabamunuge J, Dagher Z, Slingerland AE, Del Rio C, Valles B, Kempner ME, Smith M, Brown J, Dey BR, El-Jawahri A, McAfee SL, Spitzer TR, Ballen KK, Sung AD, Dalton TE, Messina JA, Dettmer K, Liebisch G, Oefner P, Taur Y, Pamer EG, Holler E, Mansour MK, van den Brink MRM, Hohmann E, Jenq RR, Chen YB. Third-party fecal microbiota transplantation following allo-HCT reconstitutes microbiome diversity. Blood Adv. 2018 Apr 10;2(7):745-753. doi: 10.1182/bloodadvances.2018017731. PMID 29592876